CLINICAL TRIAL: NCT02821273
Title: Modified INSURE vs INSURE in Preterm Infants With Respiratory Distress Syndrome: A Randomized Controlled Trials
Brief Title: Surfactant Administration in Preterm Infants
Acronym: surfactant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Fang Wu, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INSURE technique
Record Dates: First submitted 2016-06-24; First posted 2016-07-01 (Estimated); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Modified INSURE Technique

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Modified INSURE (Experimental): Modified INSURE is intubation-surfactant-X-ray relieved-extubation. Extubation and noninvasive ventilation is used after the X-ray relieving.
  Interventions: Other: Modified INSURE technique
- INSURE (Active Comparator): INSURE technique meas surfactant administration through intubation-surfactant-extubation. And noninvasive ventilation is immediately used after surfactant.
  Interventions: Other: INSURE technique

INTERVENTIONS:
Other: Modified INSURE technique — modified INSURE means intubation-surfactant-X-ray relieved-extubation. Extubation and noninvasive ventilation is used after the X-ray relieving.
  Arms: Modified INSURE
Other: INSURE technique — INSURE means intubation-surfactant-extubation. Extubation and noninvasive ventilation is used after surfactant administration.
  Arms: INSURE

SUMMARY:
In preterm infants with respiratory distress syndrome, mechanical ventilation is related to increased risk of death and complications. Surfactant is an important methods to reduce mortality and intubation rates. INSURE technique is a standard method to administrate surfactant. However, several preterm infants need two or more surfactant, and therefore one more intubation is needed. How to reduce the times of intubation is an challenges for neonatologists.

DETAILED DESCRIPTION:
INSURE technique meas surfactant administration through intubation-surfactant-extubation. And noninvasive ventilation is immediately used after surfactant.

The differences of modified INSURE compared with INSURE is intubation-surfactant-X-ray relieved-extubation. Extubation and noninvasive ventilation is used after the X-ray relieving.

ELIGIBILITY:
Inclusion Criteria:

* All preterm infants with respiratory distress syndrome

Exclusion Criteria:

* congenital abnormalities or refuse the trials

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
intubation rate | 100-days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pediatrics,Daping Hospital, Chongqing, Chongqing Municipality, China